CLINICAL TRIAL: NCT00297882
Title: Phase III Clinical Trials of Artemisinin-based Combination Therapy in Cameroon
Brief Title: Artemisinin-Based Combination Therapy: Clinical Trials in Cameroon
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: University of Yaounde (Other); Cameroon Baptist Convention Health (Other)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ITCRVG46
Record Dates: First submitted 2006-02-28; First posted 2006-03-01 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Malaria
Keywords: Efficacy; Safety; Children; Cameroon
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 Artemether-Lumefantrine (AL) (Active Comparator): Study group 1. Subjects in this group received treatment with Artemether-Lumefantrine. Children received 2 mg/kg Artemether and 12 mg/kg Lumefrantrine with milk twice daily (or every 12 hours for 3 days.
  Interventions: Drug: 1. Artemether-Lumefantrine (AL)
- 2 Amodiaquine-Artesunate (AQ-AS) (Active Comparator): Study group 2. Subjects in this group received treatment with Amodiaquine-Artesunate. Children received a co-administered combination of 30 mg/kg Amodiaquine (AQ) plus 4 mg/kg Artesunate (AS) daily for 3 days.
  Interventions: Drug: 2. Amodiaquine-Artesunate (AQ-AS)

INTERVENTIONS:
Drug: 1. Artemether-Lumefantrine (AL) — Artemether-Lumefantrine(Co-Artem)=Artemether, 2mg/kg x 2(12h apart) and Lumefantrine, 12mg/kgx2 (12h apart).
  Other Names: CoArtem
  Arms: 1 Artemether-Lumefantrine (AL)
Drug: 2. Amodiaquine-Artesunate (AQ-AS) — Amodiaquine-Artesunate (0H),D1(24H),D2(48H)= Artesunate 4mg/kg and Amodiaquine at 10mg/kg
  Other Names: Arsucam
  Arms: 2 Amodiaquine-Artesunate (AQ-AS)

SUMMARY:
This proposal aims to evaluate the safety and efficacy of artemisinin-based anti-malaria combination drugs (ACTs) for the treatment of children aged 6-120 months in different locations in Cameroon. Randomized clinical trials will provide local data on the safety of the test drugs, and on putative marker mutations of the development of resistance to ACT. The study will involve three centers, namely, Banso (Guinea-Savannah region), Limbe(Littoral Forest), and Garoua(Sahel-Savannah). The trial will compare the efficacy and safety of Amodiaquine(AQ)-Artesunate(Art) with Coartem®(Artemether-Lumefantrine). Drug efficacy will be determined using a WHO standardized 28-day protocol. Safety will be monitored through clinical examination and biochemical and hematological indices. Molecular markers of artemisinin resistance will be investigated by molecular sequencing and comparison of parasite profiles of the PfATP6 gene in drug failure cases, . Recrudescences or re-infections will be assessed by analysis of the msp1 and msp2 genes. The impact of these combinations on generation of gametocytes will be determined from gametocyte carriage rates measured by microscopy.

DETAILED DESCRIPTION:
* Outpatients will be screened for malaria by blood film examination
* Malaria-positive children will be examined by the physician for inclusion or exclusion(see below)
* Informed consent will be sought from the guardians of potential patients
* Patients or guardians will be interviewed and a case record form completed
* Patients will be randomized into one of the two arms in the ratio 4:1 AQ/Art: CoArtem and issued a study card
* Filter paper and 5ml venous blood samples will be collected
* Patients will be hospitalised for three days to allow completion of therapy under observation
* The patient will be asked to return on days 7, 14 and 28 for assessment of clearance or recrudescence of parasites
* Patient will be examined for parasites and evaluated for early treatment failure (ETF), late treatment failure (LTF), late parasitological failure (LPF) or adequate clinical and parasitological response.(ACPR).
* If a patient does not appear for follow up, a community health worker will try to trace them and will collect blood onto filter paper and a microscope slide should the patient have a temperature ≥ 37.5°C
* Patients whose parents opt out of the study will be administered quinine sulphate if parasitaemic
* Filter paper samples will be air dried and stored with dessicant until required.
* Whole blood samples collected into citrate as anticoagulant will be processed for plasma, aliquoted into 300µl lots and stored at -70°C.
* Patient information will be entered at the close of each day into laptops and collectively sent to Yaounde at the end of the first month of study and thereafter at the end of each week, along with the hard copies of the case report forms.
* Analysis will be performed on the samples within three months of collection for molecular markers of resistance, genetic structure of parasites and for blood drug levels of medications used in the trial

ELIGIBILITY:
Inclusion criteria:

* children aged 6-120 months;
* axillary temperature ≥ 37.5°C and/or history of fever within past 24 hours;
* P. falciparum asexual parasitemia between 1000 and 100000/µl;
* ability to attend follow-up visits.

Exclusion criteria:

* co-infections;
* underlying chronic disease;
* severe malaria as indicated by hyperparasitemia, severe anemia (PCV 15%, Hb 5g/ml), respiratory distress, inability to drink, persistent vomiting in past 24 hours;
* recent history of multiple convulsions;
* jaundice;
* the inability to stand or sit;
* history of allergy to study drugs.

Ages: 6 Months to 120 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 816 (Actual)
Dates: Start 2006-07; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilfred F Mbacham, ScD, Principal Investigator — University of Yaounde

IPD SHARING:
Plan to Share IPD: Yes
Database available on request of Prof Wilfred Mbacham wfmbacham@yahoo.com
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 2013 and for 10 years
Access Criteria: Database available on reqeust of Prof Wilfred Mbacham wfmbacham@yahoo.com
URL: https://www.gatesmalariapartnership.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight hundred and sixteen children aged 6-120 months with uncomplicated falciparum malaria were studied in three ecological different regions of Cameroon - Mutengene (Littoral equatorial forest), Bangolan (Rice farming guinea-savanna) and Garoua (Guinea-savannah).
Groups:
- 1 Artemether-Lumefantrine: Drug: Artemether-Lumefantrine, Artemether-Lumefantrine(Co-Artem) =Artemether, 2mg/kg x 2 (12H apart)/Lumefantrine, 12mg/kgx2 (12H apart).
  Other Names: • CoArtem,
- 2 Amodiaquine- Artesunate: Drug: Amodiaquine-Artesunate Amodiaquine-Artemether - administration D0 (0H), D1 (24H), D2 (48H)- Artesunate 4mg/kg & Amodiaquine at 10mg/kg Other Names: • Arsucam
Period: Day 14
Arm/Group | 1 Artemether-Lumefantrine | 2 Amodiaquine- Artesunate
Started | 204 | 612
Completed | 192 | 563
Not Completed | 12 | 49
Not completed — Lack of Efficacy | 12 | 49
Period: Day 28
Arm/Group | 1 Artemether-Lumefantrine | 2 Amodiaquine- Artesunate
Started | 192 | 563
Completed | 176 | 540
Not Completed | 16 | 23
Not completed — Lost to Follow-up | 13 | 23
Not completed — Lack of Efficacy | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 Artemether-Lumefantrine; 2 Amodiaquine-Artemether: Artemether-Lumefantrine , Amodiaquine-Artesunate: 1 Artemether-Lumefantrine(Co-Artem)=Artemether, 2mg/kg x 2(12h apart) and Lumefantrine, 12mg/kgx2 (12h apart).
  2 Amodiaquine-ArtemetherD0(0H),D1(24H),D2(48H)- Artesunate 4mg/kg and Amodiaquine at 10mg/kg
- Total: Total of all reporting groups
Arm/Group | 1 Artemether-Lumefantrine | 2 Amodiaquine-Artemether | Total
Number analyzed (Participants) | 204 | 612 | 816
Age, Continuous [Mean (Standard Deviation); unit: months] — Population: 100 did not complete the trial including 4 deaths
  months | 52.87 (28.4) | 50.77 (27.33) | 51.82 (27.87)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 100 did not complete trial, including 4 deaths
  Participants
    Female | 104 | 302 | 406
    Male | 100 | 310 | 410
Region of Enrollment [Number; unit: participants]
  Cameroon | 204 | 612 | 816

OUTCOME MEASURES:

1. Primary Outcome: Cure Rate on Day 28
Description: To evaluate the safety and antimalarial efficacy of two drug combinations: Artemether-Lumefantrine (AL) and Amodiaquine-Artesunate (AQ - AS) in Camaroonian patients in Mutengene, Bangolan and Garoua
Time Frame: Day 0 - 28
Population: Children aged 6 months-10 years in different locations in Cameroon.
Measure: Count of Participants; unit: Participants
Groups:
- 1 Artemether-Lumefantrine AL: 1Artemether-Lumefantrine(Co-Artem)=Artemether, 2mg/kg x 2(12h apart) and Lumefantrine, 12mg/kgx2 (12h apart).
- 2 Amodiaquine-Artesunate AQ-AS: 2 Amodiaquine-Artesunate 4mg/kg and Amodiaquine at 10mg/kg
Arm/Group | 1 Artemether-Lumefantrine AL | 2 Amodiaquine-Artesunate AQ-AS
Number analyzed (Participants) | 204 | 612
Participants | 197 | 603
Statistical Analysis 1: Comparison: 1 Artemether-Lumefantrine AL vs 2 Amodiaquine-Artesunate AQ-AS; Sample Size will be determined by N = {[(Zα/2)/E]*2}pq where Where: n=sample size; Zα/2= Z value of a two-tailed test with 95% confidence level=1.96; p represents cure rate, q=1-p, which represents treatment failure rate of; E=precision of 5%; Test type: Non-Inferiority — Non-inferiority of AQ-AS compared to AL was assessed by constructing a one-sided, lower limit asymptotic 97.5% CI on the difference of polymerase chain reaction (PCR)-corrected cure rates of AQ-AS when compared to AL. Non-inferiority was declared if the lower limit of the CI was greater than -10% for AQ-AS; p > 0.05, t-test, 2 sided

2. Secondary Outcome: Cure Rate Day 14
Description: To evaluate antimalarial efficacy of AL and AQ-AS on day 14 post-treatment
Time Frame: Day 0-14
Measure: Count of Participants; unit: Participants
Groups:
- 1 Artemether-Lumefantrine: 1Artemether-Lumefantrine(Co-Artem)=Artemether, 2mg/kg x 2(12h apart) and Lumefantrine, 12mg/kgx2 (12h apart).
- 2 Amodiaquine-Artesunate: 2 Amodiaquine-Artesunate 4mg/kg and Amodiaquine at 10mg/kg every day for 3 days
Arm/Group | 1 Artemether-Lumefantrine | 2 Amodiaquine-Artesunate
Number analyzed (Participants) | 204 | 612
Participants | 192 | 563
Statistical Analysis 1: Comparison: 1 Artemether-Lumefantrine vs 2 Amodiaquine-Artesunate; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p > 0.05, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 28 days following treatment.
Groups:
- 1 Artemether-Lumefantine (AL): Study group 1. Subjects in this group received treatment with Artemether-Lumefantrine. Children received 2 mg/kg Artemether and 12 mg/kg Lumefrantrine with milk twice daily (or every 12 hours for 3 days.
Arm/Group | 1 Artemether-Lumefantine (AL) | 2 Amodiaquine-Artesunate (AQ-AS)
All-Cause Mortality (participants affected / at risk) | 2/204 | 2/612
Serious Adverse Events (participants affected / at risk) | 6/204 | 3/612
Other Adverse Events (participants affected / at risk) | 105/204 | 272/612
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Artemether-Lumefantine (AL) (N=204) | 2 Amodiaquine-Artesunate (AQ-AS) (N=612)
Event leading to death (Infections and infestations) | 2 (2) | 2 (2) — Malaria
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Blackwater fever (Infections and infestations) | 1 (1) | 0 (0)
Hemoglobinuria (Hepatobiliary disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Artemether-Lumefantine (AL) (N=204) | 2 Amodiaquine-Artesunate (AQ-AS) (N=612)
Leucopenia (Blood and lymphatic system disorders) | 53 (53) | 139 (139)
Lymphopenia (Blood and lymphatic system disorders) | 29 (29) | 93 (93)
Neutropenia (Blood and lymphatic system disorders) | 15 (15) | 20 (20)
Thrombocytopenia (Blood and lymphatic system disorders) | 9 (9) | 20 (20)
Abdominal pain (Gastrointestinal disorders) | 25 (25) | 63 (63)
Anorexia (Gastrointestinal disorders) | 31 (31) | 123 (123)
Itching (Skin and subcutaneous tissue disorders) | 3 (3) | 12 (12)
Cuteneous eruptions (Skin and subcutaneous tissue disorders) | 3 (3) | 21 (21)
Diarrhea (Gastrointestinal disorders) | 32 (32) | 21 (21)
Vomiting (Gastrointestinal disorders) | 15 (15) | 23 (23)

LIMITATIONS AND CAVEATS:
There were no limitations or caveats that prevented completion of the trial as planned

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No